CLINICAL TRIAL: NCT05973682
Title: Effects of Post Isometric Relaxation With Scapular Stabilization Exercises on Pain, Range of Motion and Disability With Levator Scapulae Syndrome
Brief Title: Effects of Post Isometric Relaxation With Scapular Stabilization Exercises
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/0127 Kainat
Record Dates: First submitted 2023-06-27; First posted 2023-08-03 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Upper Cross Syndrome
Keywords: Neck muscles; Neck Pain; levator scapulae; Range of Motion
MeSH Terms: conditions — Oculocerebral hypopigmentation syndrome type Preus; Neck Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: post isometric relaxation and ConVentional treatment. (Experimental): Post Isometric Relaxation: The term refers to the effect of subsequent relaxation experienced by a muscle or group of muscles, after brief periods during which an isometric contraction has been performed. Post isometric relaxation technique was applied to levator scapulae for 5 repetition using 20% of maximal isometric contraction for 7-10 sec. with complete relaxation of all element, the stretch is maintained for 30 sec.
  Interventions: Other: Post-isometric relaxation and Conventional treatment; Other: Conventional Physical Therapy
- Group B: Conventional treatment (Active Comparator): hot pack and TENS at neck area for 10 mint upper trapezius, levator scapulae and pectoralis stretching 3 times with 30-second hold. static stretching exercises, two sessions per week for 3 weeks were given to each patient
  Interventions: Other: Conventional Physical Therapy

INTERVENTIONS:
Other: Post-isometric relaxation and Conventional treatment — The term refers to the effect of subsequent relaxation experienced by a muscle or group of muscles, after brief periods during which an isometric contraction has been performed. Post isometric relaxation technique was applied to levator scapulae for 5 repetition using 20% of maximal isometric contraction for 7-10 sec. with complete relaxation of all element, the stretch is maintained for 30 sec.
  + hot pack and TENS at neck area for 10 mint upper trapezius, levator scapulae and pectoralis stretching 3 times with 30 second hold. static stretching exercises two sessions per week for 3 weeks were given to each patient
  Arms: Group A: post isometric relaxation and ConVentional treatment.
Other: Conventional Physical Therapy — Conventional Physical Therapy; hot pack and TENS at neck area for 10 mint upper trapezius, levator scapulae and pectoralis stretching 3 times with 30-second hold. static stretching exercises, two sessions per week for 3 weeks were given to each patient

SUMMARY:
The levator scapulae is an important postural muscle that tends to shorten or become tight because of overactivity and bad posture, leading to neck and shoulder pain. Levator scapulae syndrome is usually caused by the poor shoulders posture as rounded shoulders as sitting at a computer hunched. It is exacerbated by sustained neck postures, neck movements or levator scapulae muscle palpation. The aim of study will be to determine the effects of post isometric relaxation with scapular stabilization exercises on pain, disability and range of motion in patients with levator scapulae syndrome.

DETAILED DESCRIPTION:
A Randomized Controlled Trial will be conducted at Tehsil Headquarter Hospital Sharqpur Shareef, Sheikhupura through consecutive sampling technique on 30 patients with levator scapulae syndrome which will be allocated using simple random sampling through sealed opaque enveloped into Group A and Group B. Group A will be treated with post isometric relaxation, scapular stabilization exercises along with baseline treatment. Group B will be treated with post isometric relaxation along with baseline treatment. Baseline treatment includes hot pack, TENS, upper trapezius stretch, levator scapular stretch and pectoralis major stretch. Both groups will come thrice per week for a total of 4 weeks. Outcome measures are NPRS, universal goniometer and NDI. Data will be analysed during SPSS software version 25. After assessing normality of data by Shapiro-Wilk test, it will be decided either parametric or non-parametric test will be used within a group or between two groups.

Keywords: Disability, Levator Scapulae, Range of Motion, Pain

ELIGIBILITY:
Inclusion Criteria:

* Both Males and females
* Age range of 18-40 years
* Neck and medial border scapular pain for at least 3months
* Examination - Increased muscle tone and tenderness at neck
* Reduced Side flexion and Rotation of neck
* Positive Levator Scapular length Test

Exclusion Criteria:

* Neuropathies
* Vertebral fractures
* Pregnancy
* Previous cognitive and functional disorders
* Traumatic neck injury
* Fibromyalgia
* cancer

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-10-05 (Actual); Primary Completion 2024-03-08 (Actual); Study Completion 2024-03-10 (Actual)

PRIMARY OUTCOMES:
Universal Goniometer (UG) | upto 4 weeks
  Universal Goniometer (UG) used to measure ROM of cervical Spine
  A goniometer is an instrument that measures the available range of motion at a joint. Physical therapists commonly use a goniometer to measure the range of motion. The therapist can use a goniometer to assess the range of motion at the initial assessment. In this study range of motion of the neck will be measured.
  The cervical spine's range of motion is approximately 80° to 90° of flexion, 70° of extension, 20° to 45° of lateral flexion, and up to 90° of rotation to both sides.
Numeric pain rate scale (NPRS) | upto 4 weeks
  The numeric pain rate scale (NPRS) measures the pain at the neck region in patients with mechanical neck pain.
  The patient's level of pain will be assessed using this scale. This scale ranges from 0 to 10. 0 indicates "no pain", and 10 indicates "worst pain. NPRS is categorized into mild, moderate and severe pain.
  Mild pain value 1 to 3 Moderate pain value 4 to 7 Severe pain value 8 to 10
Neck Disability index (NDI) | upto 4 weeks
  Neck Disability index (NDI) measures the disability of the neck region in patients with mechanical pain.
  NDI questionnaire will be used to assess disability. It comprises 10 items; 7 related to daily living activities, 2 related to pain and 1 to concentration. Each item is scored from 0 to 5. The total score is a percentage, with higher scores related to more significant disability.
  0 to 4 = no disability 5 to 14 = mild 15 to 24 = moderate 25 to 34 = severe Above 34 = complete

CONTACTS AND LOCATIONS:
Overall Officials: Samrood Akram, Mphil, Principal Investigator — Riphah International University,Lahore
Locations (1):
- Tehsil Headquarter Hospital Sharqpur Shareef, Sheikhupura, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mahmoud NF, Hassan KA, Abdelmajeed SF, Moustafa IM, Silva AG. The Relationship Between Forward Head Posture and Neck Pain: a Systematic Review and Meta-Analysis. Curr Rev Musculoskelet Med. 2019 Dec;12(4):562-577. doi: 10.1007/s12178-019-09594-y. PMID 31773477
- [Background] Masaracchio M, Kirker K, States R, Hanney WJ, Liu X, Kolber M. Thoracic spine manipulation for the management of mechanical neck pain: A systematic review and meta-analysis. PLoS One. 2019 Feb 13;14(2):e0211877. doi: 10.1371/journal.pone.0211877. eCollection 2019. PMID 30759118
- [Background] Mendes-Fernandes T, Puente-Gonzalez AS, Marquez-Vera MA, Vila-Cha C, Mendez-Sanchez R. Effects of Global Postural Reeducation versus Specific Therapeutic Neck Exercises on Pain, Disability, Postural Control, and Neuromuscular Efficiency in Women with Chronic Nonspecific Neck Pain: Study Protocol for a Randomized, Parallel, Clinical Trial. Int J Environ Res Public Health. 2021 Oct 12;18(20):10704. doi: 10.3390/ijerph182010704. PMID 34682453
- [Background] Gonzalez-Rueda V, Hidalgo-Garcia C, Rodriguez-Sanz J, Bueno-Gracia E, Perez-Bellmunt A, Rodriguez-Rubio PR, Lopez-de-Celis C. Does Upper Cervical Manual Therapy Provide Additional Benefit in Disability and Mobility over a Physiotherapy Primary Care Program for Chronic Cervicalgia? A Randomized Controlled Trial. Int J Environ Res Public Health. 2020 Nov 11;17(22):8334. doi: 10.3390/ijerph17228334. PMID 33187167
- [Background] Henry JP, Munakomi S. Anatomy, Head and Neck, Levator Scapulae Muscles. 2023 Aug 28. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK553120/ PMID 31971759
- [Background] Pecos-Martin D, Ponce-Castro MJ, Jimenez-Rejano JJ, Nunez-Nagy S, Calvo-Lobo C, Gallego-Izquierdo T. Immediate effects of variable durations of pressure release technique on latent myofascial trigger points of the levator scapulae: a double-blinded randomised clinical trial. Acupunct Med. 2019 Jun;37(3):141-150. doi: 10.1136/acupmed-2018-011738. Epub 2019 May 7. PMID 31060367